CLINICAL TRIAL: NCT05101954
Title: A Comparative Study Between the Effect of Platelet-rich Fibrin and Concentrated Growth Factors on Osseointegration of Immediate Implants (a Randomized Clinical Trial)
Brief Title: Platelet Rich Fibrin and Concentrated Growth Factors on Osseointegration of Immediate Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRF_GF_2019/2020
Record Dates: First submitted 2021-10-20; First posted 2021-11-01 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Tooth Extraction; Dental Implants

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental)
  Interventions: Procedure: Concentrated Growth Factors (CGF)
- Group B (Active Comparator)
  Interventions: Procedure: Platelet-Rich Fibrin (PRF)

INTERVENTIONS:
Procedure: Concentrated Growth Factors (CGF) — Concentrated Growth Factors membrane will be laid in the implant cavity. Bone graft material will be applied to fill the empty parts of the socket.
  Arms: Group A
Procedure: Platelet-Rich Fibrin (PRF) — Platelet-Rich Fibrin (PRF) membrane will be laid in the implant cavity. Bone graft material will be applied to fill the empty parts of the socket.
  Arms: Group B

SUMMARY:
This study will involve 14 patients with mandibular premolars indicated for extraction and immediate replacement. The patients will be randomly allocated into two groups and each patient will receive one implant. In Group A, a CGF membrane will be laid in the implant cavity. While in Group B, a PRF membrane will be laid in the implant cavity. Bone graft material will be applied to fill the empty parts of the socket.

Resonance frequency measurement will be done using the OSTELL device intraoperatively, at the 1st week and after 3 months. Cone-beam computed tomography will be done preoperatively, immediately following surgery, and after 3 months

ELIGIBILITY:
Inclusion Criteria:

* Cooperative patients with good oral hygiene.
* Patients having a history of mandibular premolars indicated for extraction and immediate replacement.

Exclusion Criteria:

* Heavy smokers.
* Parafunctional occlusal habits.
* Uncontrolled diabetes.
* History of chemotherapy or radiotherapy.
* Hematological disorders that prevent either implantation or centrifugation.
* Pregnancy.
* The nee¬d for additional augmentation or previous augmentation of the same region.
* Chronic periapical pathology

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-08-17 (Actual); Study Completion 2021-08-17 (Actual)

PRIMARY OUTCOMES:
Change in implant stability | immediately, at 1 week, at 3 months
  Osstell instrument (Integration Diagnostics, Goteborg, Sweden) with Smartpeg™ (Integration Diagnostics, Goteborg, Sweden), a transducer suitable for implants will be used to assess stability of implants by RFA. ISQ (implant stability quotient) will be obtained from the measurement results. During measurement, the Smartpeg™ will be placed over the location of implant prosthesis and the Osstell probe will be approximated to it from the buccal, palatal, mesial and distal aspects of the implant giving four ISQ values. A mean ISQ for each implant is then calculated by averaging the four values. The ISQ values of the implants will be measured during the operation, at the first week and three months after the operation.
Change in Bone density | immediately, after 3 months
  The Patients will be asked to do CBCT immediately after surgery and after 3 months
Change in bone formation | immediately, after 3 months
  Amount of bone formed buccal and lingual to the implant will be assessed using CBCT
Marginal bone loss | after 3 months
  it will be assessed using CBCT

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Faculty of Dentistry, Alexandria, Egypt